CLINICAL TRIAL: NCT06456814
Title: Epidemiological Insights Into the Formation, Progression, and Rupture of Aneurysms: A Retrospective, Multi-Center Hospital-Based Study in China
Brief Title: Epidemiological Insights Into the Formation, Progression, and Rupture of Intracranial Aneurysms: A Retrospective, Multi-Center Hospital-Based Study in China
Status: Recruiting | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Collaborators: Beijing Tiantan Hospital (Other); Guangdong Provincial People's Hospital (Other); First Affiliated Hospital of Chongqing Medical University (Other); The Affiliated Hospital Of Southwest Medical University (Other)
Responsible Party: Principal Investigator, Duan Chuanzhi, Chief physican; Professor, Zhujiang Hospital
Other Study IDs: NCT20240606IA
Record Dates: First submitted 2024-06-07; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Intracranial Aneurysm; Subarachnoid Hemorrhage, Aneurysmal; Cerebral Aneurysm; Brain Aneurysm
Keywords: Intracranial aneurysm; Clinical epidemiology; Exposures
MeSH Terms: conditions — Intracranial Aneurysm; Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a retrospective, hospital-based and multi-center study aiming at investigating the potential exposures associated with the formation, progression, and rupture of intracranial aneurysms in Chinese population.

DETAILED DESCRIPTION:
A striking conflict exists between the fatal rupture of intracranial aneurysms (IA) and the passive approach to detecting IA through cerebrovascular examinations. This is attributed to a limited understanding of risk factors for IA incidence and the resulting lack of cost-effective IA screening.

This study aims to gain epidemiological insights into the exposures associated with the risk of IA incidence, including formation, progression, and rupture in the Chinese population. It integrates multi-modal data based on large-scale electronic medical records from high-volume stroke centers across China to investigate potential associations between various exposures and IA incidence.

Patients with anonymous and unique IDs were screened for the presence of IA by formal readings from digital subtraction angiography (DSA), cranial computed tomography angiography (CTA), or magnetic resonance angiography (MRA) conducted by two radiologists, which were then confirmed by two treating neurosurgeons using the raw images. Using natural language processing in conjunction with medical records and multi-modal data, patient exposures were extracted and assumed to be absent if no documentation was found across the databases.

Through a series of retrospective analyses, we aim to identify the exposures associated with IA incidence as much as possible to gather valuable insights for future prospective research.

ELIGIBILITY:
Inclusion Criteria:

1. IA diagnosis (ruptured or unruptured) or exclusion by digital subtractive angiography (DSA) or by cranial computed tomography angiography (CTA) / magnetic resonance angiography (MRA);
2. Aged ≥ 18 and ≤ 18 years old;
3. With complete demographic data including age and sex;
4. With medical record archiving officially.

Exclusion Criteria:

1. Missing data of age, sex or hypertensive status;
2. Age <18 or >80 years;
3. Pregnancy;
4. With a history of intracranial arteriovenous malformation, Moyamoya, polycystic kidney disease, Ehlers-Danlos syndrome, Gronblad-Strandberg syndrome, or Marfan syndrome;
5. Suspicion for dissecting or mycotic aneurysms or aneurysm-like lesions that were indistinguishable from the infundibulum, fenestration, dilation, or atherosclerotic remodeling on structural imaging scans.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population underwent cerebrovascular examinations, with the majority conducted in clinical settings and the minority for health screening purposes, sourced from real-world electronic medical record databases.
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Intracranial aneurysm | 2010.01.01-2024.06.01
  The presence or absence of IAs detected by digital subtractive angiography or by cranial computed tomography angiography / magnetic resonance angiography.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhujiang Hospital, Guangzhou, China

REFERENCES:
- [Derived] Lin J, Feng X, Wen Z, Huang C, Huang M, Huang J, Ge R, Xu A, Ma G, Shi H, Hu Y, Yuan H, Li C, Yi R, Jin Y, Liang S, Zhang X, Li X, Duan C. Association between triglyceride-glucose index and intracranial aneurysm rupture: findings from a retrospective study. Neurosurg Rev. 2025 Jun 21;48(1):521. doi: 10.1007/s10143-025-03680-1. PMID 40542179